CLINICAL TRIAL: NCT03769402
Title: The Influence of Citric Acid Bone Surface Etching and Bone Substitute Intra-osseous Defect Fill on Crevicular Fluid BMP-2 Release Profile (Randomized Clinical Trial)
Brief Title: The Influence of Citric Acid Bone Surface Etching and Bone Defect Fill on GCF BMP-2 Release Profile
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Moustafa Mukhtar, Teaching assistant, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 52-376
Record Dates: First submitted 2018-12-06; First posted 2018-12-07 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Intrabony Periodontal Defect
MeSH Terms: interventions — Citric Acid

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Citric acid (Active Comparator): Citric acid PH1 and concentration 50% was used for 30 seconds on bone surface before washing it off and filling the defect with xenograft
  Interventions: Drug: Citric acid
- Control (Placebo Comparator): Control test
  Interventions: Drug: Control Test

INTERVENTIONS:
Drug: Citric acid — Citric acid ph1, 50% concentration solution
  Arms: Citric acid
Drug: Control Test — Control group, xenograft was used to fill infrabony defects without treating bone surface
  Other Names: Control
  Arms: Control

SUMMARY:
This study evaluates the effect of citric acid on bone surface of infrabony defects when used for 30 seconds at ph 1 and 50% concentration before the application of bovine derived xenograft to fill the defect, Bone Morphogenic protein 2 (BMP-2) marker was evaluated in 5 different days during the first month after surgery and clinical and radiographic parameters were reassessed after 6 months

DETAILED DESCRIPTION:
Citric acid have been widely used to treat root surfaces of periodontally affected teeth in order to render it biologically suitable for fibroblast reattachment. however, systematic reviews showed no clinical significance when it was used as a root surface conditioner. Recently it was found in experimental studies that when citric acid was used on bone surface for a brief period, it increased bone formation and improved consolidation of grafted bone to bone bed. In this study infrabony defects were treated with citric acid PH 1 and 50% concentration for 30 seconds before washing it off and then application of bovine derived xenograft was done to fill the defect. BMP-2 marker was evaluated at days 1,3,7,14 and 30 by taking a sample using perio-paper from the gingival crevicular fluid (GCF) and clinical and radiographic parameters were taken after 6 months of follow-up

ELIGIBILITY:
Inclusion Criteria:

* Both genders aged between 32-60 years.
* Selected patient with a single site of:

  1. Two walled or three walled infra-bony defect.
  2. The bone defect should be at least 3 mm in depth from the crest of the alveolar bone to the base of the defect.
  3. Pocket depth of more than or equal to 5 mm.
  4. Clinical attachment loss equal or more than 3mm
* Patients ready to comply with oral hygiene measures.

Exclusion Criteria:

* Any systemic disease that contra-indicates periodontal surgery or may affect healing.
* Smokers
* Pregnant females
* Drug abusers

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Bone Morphogenic protein 2 | 1 day
  The level of Bone morphogenic protein 2 was measured in the gingival crevicular fluid using a perio-paper then the marker level was determined using an Enzyme linked immunosorbent kit (ELISA kit)
Bone Morphogenic protein 2 | 3 days
  The level of Bone morphogenic protein 2 was measured in the gingival crevicular fluid using a perio-paper then the marker level was determined using an Enzyme linked immunosorbent kit (ELISA kit)
Bone Morphogenic protein 2 | 7 days
  The level of Bone morphogenic protein 2 was measured in the gingival crevicular fluid using a perio-paper then the marker level was determined using an Enzyme linked immunosorbent kit (ELISA kit)
Bone Morphogenic protein 2 | 14 days
  The level of Bone morphogenic protein 2 was measured in the gingival crevicular fluid using a perio-paper then the marker level was determined using an Enzyme linked immunosorbent kit (ELISA kit)
Bone Morphogenic protein 2 | 30 days
  The level of Bone morphogenic protein 2 was measured in the gingival crevicular fluid using a perio-paper then the marker level was determined using an Enzyme linked immunosorbent kit (ELISA kit)

SECONDARY OUTCOMES:
Gingival Index | 6 months
  Estimation of the degree of gingival inflammation was done according to Loe where scores were given between 0-3 (0=no inflammation and 3=severe inflammation)
Plaque index | 6 months
  Estimation of the amount of dental plaque according to Silness & Loe where scores were given between 0-3 (0=no plaque and 3=presence of abundant plaque)
Probing depth | 6 months
  Estimation was done by measuring the depth from the gingival margin to the base of the periodontal pocket using a UNC-15 periodontal probe
Clinical attachment level | 6 months
  Estimation was done by measuring the distance from the cemento-enamel junction to the base of the pocket using a UNC-15 periodontal probe
Radiographic bone fill | 6 months
  Estimation was done by taking a linear measurement using RVG system from the baseline defect till the alveolar bone crest